CLINICAL TRIAL: NCT03876457
Title: SELECT2: A Randomized Controlled Trial to Optimize Patient's Selection for Endovascular Treatment in Acute Ischemic Stroke
Acronym: SELECT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Stryker Neurovascular (Industry); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Amrou Sarraj, Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G180275, Pro00056862
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Ischemic stroke; Large vessel occlusion; Endovascular thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endovascular Thrombectomy plus Medical Management (Experimental)
  Interventions: Device: Endovascular Thrombectomy; Other: Medical Management
- Medical Management (Active Comparator)
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: Endovascular Thrombectomy — Patients randomized to endovascular thrombectomy arm will receive thrombectomy plus medical management. They will be treated with thrombectomy devices (stent-retrievers or aspiration devices) currently cleared by the FDA for thrombus removal in patients experiencing an acute stroke within 24 hours of symptom onset. The devices which will be used are FDA-approved stent retrievers: the Trevo Retriever, the Solitaire Revascularization Device, EmboTrap Revascularization Device and Tigertriever Revascularization Device; and/or the aspiration devices approved by the FDA (e.g. MicroVention SOFIA Catheter, and the Penumbra thrombectomy system). The choice of thrombectomy method, primary approach/technique, whether primary aspiration or primary stent-retriever with or without aspiration, will be left up to the interventionalist, with any of the FDA-approved devices approved in the study protocol or a combination of them.
  Arms: Endovascular Thrombectomy plus Medical Management
Other: Medical Management — Patients will receive standard AHA guideline-directed medical therapy, which will include IV thrombolytic therapy available for use according to practice guidelines in patients presenting within the first 3 hours from last-seen-normal and meeting other FDA label criteria, or up to 4.5 hours from last-seen-normal and meeting other AHA guidelines. For non-thrombolysis treated patients, this will include aspirin 325 mg on day 1 followed by aspirin 81 mg or 325 mg thereafter, which will be determined by treating physician and standard deep venous thrombosis prevention therapy. Intravenous anticoagulation and dual anti-platelet therapy will be discouraged without clear documented reasoning. Post-thrombolysis patients will be treated based on standard study site protocols for these patients.

SUMMARY:
SELECT 2 evaluates the efficacy and safety of endovascular thrombectomy compared to medical management alone in acute ischemic stroke patients due to a large vessel occlusion in the distal ICA and MCA M1 who have large core on either CT (ASPECTS: 3-5) or advanced perfusion imaging ([rCBF<30%] on CTP or [ADC<620] on MRI: ≥50cc) or both and are treated within 0-24 hours from last known well.

DETAILED DESCRIPTION:
SELECT 2 is a prospective, phase III randomized, international, multicenter, assessor-blinded controlled trial evaluating the efficacy and safety of thrombectomy in patients with large core on either CT or advanced perfusion imaging treated within 0-24 hours from last known well.

Patients with the final diagnosis of an acute ischemic stroke due to a large vessel occlusion in the distal ICA and MCA M1 who have large core on either CT (ASPECTS: 3-5) or advanced perfusion imaging ([rCBF<30%] on CTP or [ADC<620] on MRI: ≥50cc) or both within 0-24 hrs from last known well will be randomized in a 1:1 ratio into thrombectomy plus medical management vs medical management alone. Patient outcomes will be measured at baseline, 24 hours post, discharge, 30 days and 90 days.

The primary endpoint is the Modified Rankin Scale (mRS) at 90 (+/- 15) days. The primary outcome is a shift on 90-day mRS. Secondary outcomes are favorable clinical outcomes: mRS score of 0-2, safety outcomes such the incidence of symptomatic intracranial hemorrhage (sICH per SITS-MOST) and Imaging endpoints such as infarct volume on MRI diffusion-weighted imaging (DWI) sequence (or CT if MRI not feasible) 24 to 72 hours after randomization. CT images will be read by iSchemaView automated ASPECTS as well as by a physician. In cases where there is disagreement, the physician reading will override the automated software reading. CT/MR perfusion images with mismatch determination will be read by iSchemaView automated RAPID software. All the images will be adjudicated by a blinded core lab at the University of Texas-Medical School at Houston.

A maximum of 560 patients will be randomized across the study sites. Covariate adaptive randomization will be used to balance the distribution of important variables. Interim analyses will be conducted at 200 and 380 patients, at which time the study may stop for efficacy or futility.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-85 years) with the final diagnosis of an acute ischemic stroke
2. NIH Stroke Scale Score (NIHSS) ≥ 6
3. Last known well to groin puncture or medical management between 0 to 24 hours
4. Pre-stroke modified Rankin Scale score (mRS) of 0-1
5. Eligible for thrombectomy or medical management
6. Signed Informed Consent obtained
7. Subject willing to comply with the protocol follow-up requirements
8. Anticipated life expectancy of at least 3 months

Specific Neuroimaging Inclusion Criteria:

1. Proven large vessel occlusion in ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial, with or without tandem MCA lesions) determined by MRA or CTA
2. Large infarct-core lesion on at least one of the following:

   * 2.1. Non-Contrast CT (ASPECTS of 3-5),
   * 2.2. CT perfusion (rCBF<30% ≥50cc),
   * 2.3. MRI-DWI (ADC<620 ≥50cc)

Exclusion Criteria:

1. Inability to undergo CT angiography and/or CT perfusion imaging (e.g., renal insufficiency, iodine/contrast allergy)
2. Co-morbid psychiatric or medical illnesses that would confound the neurological assessments
3. Treatment with thrombolytic agent beyond 4.5 hours from last known well
4. Treated with thrombolytic agent 3-4.5 hours after last known well AND any of the following:

   * 1) age >80,
   * 2) current anticoagulant use,
   * 3) history of diabetes AND prior stroke,
   * 4) NIHSS >25,
   * 5) ischemic involvement of > 1/3 MCA territory
5. Current participation in another investigational drug or device study.

Neuroimaging Exclusion Criteria

1. Patients who have both ASPECTS of 6-10 on non-contrast CT AND core volume <50 cc on perfusion imaging
2. Patients with very large core on non-contrast CT i.e. ASPECTS ≤ 2
3. Evidence of intracranial tumor (except small meningioma), acute intracranial hemorrhage, neoplasm, or arteriovenous malformation
4. A significant mass effect with midline shift
5. Evidence of internal carotid artery dissection that is flow limiting or aortic dissection
6. Intracranial stent implanted in the same vascular territory that precludes the safe deployment/removal of the neurothrombectomy device
7. Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion).
8. Signs of established infarct and large area of cerebral edema on non-contrast CT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrou Sarraj, MD, Principal Investigator — Case Western Reserve University - University Hospitals Cleveland Medical Center; (Australia and Oceania) Bruce CV Campbell, MBBS PhD, Principal Investigator — Melbourne Health; (Europe) Marc Ribo, MD, Principal Investigator — Vall d'Hebron University Hospital, Barcelona
Locations (31):
- United States (19):
  - Kaiser Permanente, Los Angeles, California
  - Baptist Health, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Ascension St. Vincent Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Westchester Medical Center, Valhalla, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital - OhioHealth, Columbus, Ohio
  - Abington Jefferson Health, Abington, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Semmes Murphey Clinic - University of Tennessee Health Science Center, Memphis, Tennessee
  - Dell Seton Medical Center at the University of Texas at Austin, Austin, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Ascension Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Liverpool Hospital - South Western Sydney Clinical School, Liverpool, New South Wales
  - The Royal Adelaide Hospital (RAH), Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
- Christchurch Hospital, Christchurch, Canterbury, New Zealand
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Universität Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarraj A, Blackburn S, Abraham MG, Hussain MS, Ortega-Gutierrez S, Chen M, Kasner SE, Churilov L, Sitton CW, Pujara DK, Sundararajan S, Hu YC, Herial NA, Budzik RF, Hicks WJ, Vora N, Arenillas JF, Alfonso ML, Ramos Araque ME, Tsai JP, Abdulrazzak MA, Kozak O, Yan B, Mitchell PJ, Cordato DJ, Manning NW, Cheung A, Hanel RA, Aghaebrahim AN, Wu TY, Portela PC, Merchan AJP, Gandhi CD, Al-Mufti F, Samaniego EA, Maali L, Qureshi A, Lechtenberg CG, Slavin S, Rosterman L, Gibson D, Wallace AN, Sahlein D, Perez de la Ossa N, Hernandez Perez M, Schaafsma JD, Blasco J, Renu A, Sangha N, Warach S, Kleinig TJ, Mullen M, Elijovich L, Shaker F, Al-Shaibi FK, Johns H, Duncan KR, Opaskar A, Popovic MJ, Altose M, Ray A, Xiong W, Sunshine J, DeGeorgia M, Nguyen TN, Fifi JT, Tjoumakaris S, Jabbour P, Pereira VM, Lansberg MG, Albers GW, Sila C, Bambakidis N, Davis S, Wechsler L, Hill MD, Grotta JC, Ribo M, Hassan AE, Campbell BC; SELECT2 Investigators. General vs Nongeneral Anesthesia for Endovascular Thrombectomy in Patients With Large Core Strokes: A Prespecified Secondary Analysis of SELECT2 Trial. Neurology. 2025 Jul 22;105(2):e213819. doi: 10.1212/WNL.0000000000213819. Epub 2025 Jun 26. PMID 40570276
- [Derived] Yogendrakumar V, Campbell BCV, Johns HT, Churilov L, Ng FC, Sitton CW, Hassan AE, Abraham MG, Ortega-Gutierrez S, Hussain MS, Chen M, Kasner SE, Sharma G, Guha P, Pujara DK, Shaker F, Lansberg MG, Wechsler LR, Nguyen TN, Fifi JT, Hill MD, Ribo M, Parsons MW, Davis SM, Grotta JC, Albers GW, Sarraj A; SELECT2 Investigators. Association of Ischemic Core Hypodensity With Thrombectomy Treatment Effect in Large Core Stroke: A Secondary Analysis of the SELECT2 Randomized Controlled Trial. Stroke. 2025 Jun;56(6):1366-1375. doi: 10.1161/STROKEAHA.124.048899. Epub 2025 Mar 28. PMID 40151939
- [Derived] Ortega-Gutierrez S, Rodriguez-Calienes A, Pujara D, Sitton C, Galecio-Castillo M, Hassan AE, Abraham MG, Chen M, Blackburn S, Kasner SE, Olalde H, Ghannam M, Hussain MS, Leira EC, Martinez-Galdamez M, Shaban A, Tsai JP, Roeder H, Gudenkauf JC, Budzik R, Vora N, Hanel RA, Aghaebrahim A, Colgan F, de Miquel MA, Gandhi CD, Al-Mufti F, Blasco J, San Roman Manzanera L, Herial NA, Manning NW, Cheung A, Kozak O, Yan B, Mitchell PJ, Ebersole K, Toth G, Gooch M, Gibson D, Sahlein DH, Amuluru K, Abdulrazzak MA, Duncan K, Defta D, Shaker F, Al-Shaibi F, Ray A, Sunshine J, Hu YC, Burkhardt JK, Mir O, Alenzi B, Kass-Hout T, Gupta R, Tjoumakaris SI, Jabbour PM, Nguyen TN, Fifi JT, Pereira VM, Bambakidis N, Hill MD, Grotta JC, Ribo M, Campbell BCV, Samaniego EA, Sarraj A. Endovascular Thrombectomy for Extracranial Internal Carotid Artery Occlusions With Large Ischemic Strokes: Insights From the SELECT2 Trial. Neurology. 2025 Feb 25;104(4):e210269. doi: 10.1212/WNL.0000000000210269. Epub 2025 Jan 27. PMID 39869840
- [Derived] Tsai JP, Nguyen TN, Pujara DK, Fifi JT, Sundararajan S, Schaafsma JD, Perez de la Ossa N, Abraham MG, Chen M, Hussain MS, Ortega-Gutierrez S, Johns HT, Duncan KR, Churilov L, Lechtenberg CG, Slavin SJ, Opaskar A, de Lera M, Lara-Rodriguez B, Quesada H, Fournier LE, Defta DM, Shaker F, Sitton CW, Sharrief AZ, Grotta JC, Hill MD, Ribo M, Hassan AE, Campbell BCV, Sila C, Tjoumakaris SI, Sarraj A; for SELECT2 Investigators. Sex-Based Differences in Endovascular Thrombectomy Outcomes for Large Ischemic Stroke: A SELECT2 Subanalysis. Stroke. 2025 Feb;56(2):294-304. doi: 10.1161/STROKEAHA.124.049307. Epub 2025 Jan 2. PMID 39744837
- [Derived] Chen H, Malhotra A, Gandhi D. Thrombectomy for Large Strokes. N Engl J Med. 2024 Jul 25;391(4):378-379. doi: 10.1056/NEJMc2406965. No abstract available. PMID 39047249
- [Derived] Sarraj A, Hill MD, Hussain MS, Abraham MG, Ortega-Gutierrez S, Chen M, Kasner SE, Churilov L, Pujara DK, Johns H, Blackburn S, Sundararajan S, Hu YC, Herial NA, Budzik RF, Hicks WJ, Arenillas JF, Tsai JP, Kozak O, Cordato DJ, Hanel RA, Wu TY, Portela PC, Gandhi CD, Al-Mufti F, Maali L, Gibson D, Perez de la Ossa N, Schaafsma JD, Blasco J, Sangha N, Warach S, Kleinig TJ, Shaker F, Sitton CW, Nguyen T, Fifi JT, Jabbour P, Furlan A, Lansberg MG, Tsivgoulis G, Sila C, Bambakidis N, Davis S, Wechsler L, Albers GW, Grotta JC, Ribo M, Campbell BC, Hassan AE; SELECT2 Investigators; SELECT2 Collaborators; Vora N, Manning NW, Cheung A, Aghaebrahim AN, Paipa Merchan AJ, Sahlein D, Requena Ruiz M, Elijovich L, Arthur A, Al-Shaibi F, Samaniego EA, Duncan KR, Opaskar A, Ray A, Xiong W, Sunshine J, DeGeorgia M, Tjoumakaris S, Mendes Pereira V; SELECT2 Collaborators. Endovascular Thrombectomy Treatment Effect in Direct vs Transferred Patients With Large Ischemic Strokes: A Prespecified Analysis of the SELECT2 Trial. JAMA Neurol. 2024 Feb 8;81(4):327-35. doi: 10.1001/jamaneurol.2024.0206. Online ahead of print. PMID 38363872
- [Derived] Sarraj A, Abraham MG, Hassan AE, Blackburn S, Kasner SE, Ortega-Gutierrez S, Hussain MS, Chen M, Johns H, Churilov L, Pujara DK, Shaker F, Maali L, Cardona Portela P, Herial NA, Gibson D, Kozak O, Arenillas JF, Yan B, Perez de la Ossa N, Sundararajan S, Hu YC, Cordato DJ, Manning NW, Hanel RA, Aghaebrahim AN, Budzik RF, Hicks WJ, Blasco J, Wu TY, Tsai JP, Schaafsma JD, Gandhi CD, Al-Mufti F, Sangha N, Warach S, Kleinig TJ, Yogendrakumar V, Ng F, Samaniego EA, Abdulrazzak MA, Parsons MW, Rahbar MH, Nguyen TN, Fifi JT, Mendes Pereira V, Lansberg MG, Albers GW, Furlan AJ, Jabbour P, Sitton CW, Sila C, Bambakidis N, Davis SM, Wechsler L, Hill MD, Grotta JC, Ribo M, Campbell BCV; SELECT2 Investigators. Endovascular thrombectomy plus medical care versus medical care alone for large ischaemic stroke: 1-year outcomes of the SELECT2 trial. Lancet. 2024 Feb 24;403(10428):731-740. doi: 10.1016/S0140-6736(24)00050-3. Epub 2024 Feb 9. PMID 38346442
- [Derived] Sarraj A, Hassan AE, Abraham MG, Ortega-Gutierrez S, Kasner SE, Hussain MS, Chen M, Churilov L, Johns H, Sitton CW, Yogendrakumar V, Ng FC, Pujara DK, Blackburn S, Sundararajan S, Hu YC, Herial NA, Arenillas JF, Tsai JP, Budzik RF, Hicks WJ, Kozak O, Yan B, Cordato DJ, Manning NW, Parsons MW, Cheung A, Hanel RA, Aghaebrahim AN, Wu TY, Portela PC, Gandhi CD, Al-Mufti F, Perez de la Ossa N, Schaafsma JD, Blasco J, Sangha N, Warach S, Kleinig TJ, Shaker F, Al Shaibi F, Toth G, Abdulrazzak MA, Sharma G, Ray A, Sunshine J, Opaskar A, Duncan KR, Xiong W, Samaniego EA, Maali L, Lechtenberg CG, Renu A, Vora N, Nguyen T, Fifi JT, Tjoumakaris SI, Jabbour P, Tsivgoulis G, Pereira VM, Lansberg MG, DeGeorgia M, Sila CA, Bambakidis N, Hill MD, Davis SM, Wechsler L, Grotta JC, Ribo M, Albers GW, Campbell BC; SELECT2 Investigators. Endovascular Thrombectomy for Large Ischemic Stroke Across Ischemic Injury and Penumbra Profiles. JAMA. 2024 Mar 5;331(9):750-763. doi: 10.1001/jama.2024.0572. PMID 38324414
- [Derived] Sarraj A, Hassan AE, Abraham MG, Ortega-Gutierrez S, Kasner SE, Hussain MS, Chen M, Blackburn S, Sitton CW, Churilov L, Sundararajan S, Hu YC, Herial NA, Jabbour P, Gibson D, Wallace AN, Arenillas JF, Tsai JP, Budzik RF, Hicks WJ, Kozak O, Yan B, Cordato DJ, Manning NW, Parsons MW, Hanel RA, Aghaebrahim AN, Wu TY, Cardona-Portela P, Perez de la Ossa N, Schaafsma JD, Blasco J, Sangha N, Warach S, Gandhi CD, Kleinig TJ, Sahlein D, Elijovich L, Tekle W, Samaniego EA, Maali L, Abdulrazzak MA, Psychogios MN, Shuaib A, Pujara DK, Shaker F, Johns H, Sharma G, Yogendrakumar V, Ng FC, Rahbar MH, Cai C, Lavori P, Hamilton S, Nguyen T, Fifi JT, Davis S, Wechsler L, Pereira VM, Lansberg MG, Hill MD, Grotta JC, Ribo M, Campbell BC, Albers GW; SELECT2 Investigators. Trial of Endovascular Thrombectomy for Large Ischemic Strokes. N Engl J Med. 2023 Apr 6;388(14):1259-1271. doi: 10.1056/NEJMoa2214403. Epub 2023 Feb 10. PMID 36762865
- [Derived] Sarraj A, Campbell BCV, Christensen S, Sitton CW, Khanpara S, Riascos RF, Pujara D, Shaker F, Sharma G, Lansberg MG, Albers GW; SELECT Investigators. Accuracy of CT Perfusion-Based Core Estimation of Follow-up Infarction: Effects of Time Since Last Known Well. Neurology. 2022 May 24;98(21):e2084-e2096. doi: 10.1212/WNL.0000000000200269. Epub 2022 Apr 21. PMID 35450966
- [Derived] Sarraj A, Hassan AE, Abraham M, Ribo M, Blackburn S, Chen M, Hussain MS, Pereira VM, Ortega-Gutierrez S, Sitton C, Lavori PW, Cai C, Rahbar M, Pujara D, Shaker F, Lansberg MG, Campbell B, Grotta JC, Albers GW; SELECT2 Investigators. A randomized controlled trial to optimize patient's selection for endovascular treatment in acute ischemic stroke (SELECT2): Study protocol. Int J Stroke. 2022 Jul;17(6):689-693. doi: 10.1177/17474930211035032. Epub 2021 Dec 15. PMID 34282987

RESULTS

PARTICIPANT FLOW:
Groups:
- Endovascular Thrombectomy Plus Medical Management: Endovascular Thrombectomy: Patients will receive thrombectomy plus medical management. Treated with thrombectomy devices (stent-retrievers or aspiration devices) currently cleared by the FDA for thrombus removal in patients experiencing an acute stroke within 24 hours of symptom onset. The devices used are FDA-approved: Trevo Retriever, the Solitaire Revascularization Device, EmboTrap Revascularization Device and Tigertriever Revascularization Device; and/or the aspiration devices approved by the FDA (e.g. MicroVention SOFIA Catheter, and the Penumbra thrombectomy system). The choice of thrombectomy method, primary approach/technique, whether primary aspiration or primary stent-retriever with/without aspiration, is left up to the interventionalist.
  Medical Management: Patients receive AHA guideline-directed medical therapy- includes IV thrombolytic therapy for use according to practice guidelines in patients presenting within the first 3 hours from last-seen-normal and meeting other FDA label criteria, or up to 4.5 hours from last-seen-normal and meeting other AHA guidelines. Non-thrombolysis treated patients: includes aspirin 325 mg on day 1, then aspirin 81 mg or 325 mg thereafter, will be determined by treating physician and standard deep venous thrombosis prevention therapy. Intravenous anticoagulation and dual anti-platelet therapy will be discouraged without clear documented reasoning. Post-thrombolysis patients will be treated based on standard study site protocols.
Period: Overall Study
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Started | 178 | 174
Completed | 177 | 171
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management | Total
Number analyzed (Participants) | 178 | 174 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.7) | 65.3 (12.6) | 65.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 74 | 145
  Male | 107 | 100 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 136 | 134 | 270
  Unknown or Not Reported | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 26 | 24 | 50
  White | 132 | 130 | 262
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Degree of Disability/Dependence as Measured by the Modified Rankin Scale (mRS) Score
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
Time Frame: 90 days
Measure: Median (95% Confidence Interval); unit: scores on a scale
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
scores on a scale | 4 [3 to 6] | 5 [4 to 6]

2. Secondary Outcome: Number of Participants That Achieved Functional Independence as Measured by a mRS Score of 0-2 at 90-day Follow-up
Description: as for outcome 1
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 171
Participants | 36 | 12

3. Secondary Outcome: Number of Participants That Achieved Independent Ambulation as Measured by a mRS Score of 0-3 at 90-day Follow-up
Description: as for outcome 1
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 171
Participants | 67 | 32

4. Secondary Outcome: Number of Patients That Suffered a Symptomatic Intracranial Hemorrhage (sICH) as Measured by the SITS-MOST Criteria
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants | 1 | 2

5. Secondary Outcome: Number of Participants With Neurological Worsening Defined as a ≥4-point Increase on the NIHSS Score Due to the Stroke Itself
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants | 44 | 27

6. Secondary Outcome: Number of Mortalities Within 90-day Follow-up
Time Frame: 90 days
Measure: Number; unit: Mortalities
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 171
Mortalities | 68 | 71

7. Secondary Outcome: Number of Procedural Complications
Description: The following were included in the complications counted:
  * Surgical site hematoma
  * Surgical site infection
  * Vascular injury (peripheral or intracranial dissection, perforation or others) caused by the endovascular procedure
Time Frame: 24 hours
Population: Patients in the medical management group did not undergo procedure so no data was collected for that group.
Measure: Number; unit: Procedural complications
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 0
Procedural complications | 30 |

8. Secondary Outcome: Successful Reperfusion in the EVT Group, Defined as Modified Thrombolysis in Cerebral Ischemia (mTICI) Grade of 2b or Higher
Time Frame: at the end of endovascular thrombectomy procedure
Population: Data was only collected for the Endovascular Thrombectomy plus Medical Management group
Measure: Number; unit: Successful reperfusions
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 0
Successful reperfusions | 142 |

9. Secondary Outcome: Discharge Location
Time Frame: day 5-7 after randomization/at discharge (whichever is later)
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants
  Discharged to home | 19 | 10
  Discharged to acute care facility | 11 | 16
  Discharged to inpatient rehab facility | 72 | 65
  Discharged to skilled nursing facility | 23 | 20
  Discharged to hospice or home hospice | 11 | 19
  Discharged to in-hospital death | 42 | 44

10. Secondary Outcome: Number of Participants That Showed Early Neurological Improvement, Defined as Improvement of ≥8 Points on NIHSS at 24 Hours of Presentation or an NIHSS of 0-1
Time Frame: 24 hours
Population: 4 participants in the Endovascular Thrombectomy plus medical management, and 1 participant in the medical management group did not have enough data available to be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 174 | 172
Participants | 20 | 13

11. Secondary Outcome: Quality of Life Score, as Measured Using NeuroQOL at 90-day Follow-up
Description: The Neurological Quality of Life score (NeuroQoL) is a patient-reported outcome measure that assesses the impact of neurological disorders on various aspects of a person's quality of life in neurological diseases and has measures developed across 17 different domains. The trial measured NeuroQoL scores for Mobility, Depression, Social and Cognitive domains. The scores provide a measure of an individual's quality of life in a given domain relative to a reference population, with a mean score of 50 and range of 0-100. A t-score of 50 indicates average quality of life, while scores above 50 indicate better-than-average quality of life and scores below 50 indicate poorer-than-average quality of life, except for depression domain - where lower scores indicate better and higher scores indicate worse quality of life.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 171
score on a scale
  Mobility domain | 35.2 [23.9 to 43.9] | 25.1 [16.5 to 33.0]
  Depression domain | 47.9 [43.1 to 54.3] | 53.6 [46.8 to 57.4]
  Social domain | 37.1 [32.7 to 42.0] | 33.5 [27.7 to 37.8]
  Cognitive domain | 41.9 [35.0 to 49.6] | 37.9 [30.9 to 42.9]

12. Secondary Outcome: The 1-year Functional Outcome, as Measured by the Modified Rankin Scale Score
Description: as for outcome 1
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
score on a scale | 5 [3 to 6] | 6 [4 to 6]

13. Secondary Outcome: Number of Participants With Functional Independence, Defined as mRS Score of 0-2 at 1-year Follow-up
Description: as for outcome 1
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 170 | 159
Participants | 40 | 9

14. Secondary Outcome: Number of Participants With Independent Ambulation, Defined as mRS Score of 0-3 at 1-year Follow-up
Description: as for outcome 1
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 170 | 159
Participants | 63 | 29

15. Secondary Outcome: Quality of Life Score, as Measured Using NeuroQOL at 1 Year Follow-up
Description: Quality of Life scores in mobility, depression,social and cognitive domains
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 170 | 159
score on a scale
  Mobility domain | 40.8 [26.2 to 48.6] | 27.2 [19.2 to 38.3]
  Depression domain | 45.3 [36.9 to 55.1] | 52.1 [49.7 to 57.4]
  Social domain | 40.6 [33.5 to 44.7] | 35 [30.5 to 41.3]
  Cognitive domain | 46 [37 to 59] | 38.9 [33 to 46]

16. Other Pre Specified Outcome: Infarct Volume on MRI DWI Sequence (or CT if MRI Not Feasible) up to 7 Days After Randomization
Description: Infarct volume on MRI DWI sequence (or CT if MRI not feasible) up to 7 days after randomization
Time Frame: Up to 7 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 174
mL | 178 [109 to 253] | 168.5 [124 to 268]

17. Other Pre Specified Outcome: Lesion Growth (Difference Between the Ischemic Core on Baseline Imaging and the Follow-up Infarct Volume)
Description: Lesion growth (difference between ischemic core on baseline imaging and the follow-up infarct volume)
Time Frame: 24 hours to 7 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 177 | 174
mL | 78 [22 to 131] | 65.5 [24 to 110]

18. Other Pre Specified Outcome: Number of Participants Who Suffered Parenchymal Hemorrhage Type 2
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants | 2 | 1

19. Other Pre Specified Outcome: Number of Participants Who Suffered a Subarachnoid Hemorrhage
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants | 4 | 0

20. Other Pre Specified Outcome: Number of Participants Who Had a Hemicraniectomy During Index Hospitalization
Time Frame: day 5-7 after randomization/at discharge (whichever is later)
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Participants | 29 | 26

21. Other Pre Specified Outcome: Length of Hospital Stay
Description: Was assessed if the patient was discharged at every follow-up visit to determine the length of the stay if the patient was not discharged at the time of previous follow-up visit.
Time Frame: Up to 90-day follow up visit
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
Number analyzed (Participants) | 178 | 174
Days | 9 [5 to 17] | 8 [5 to 13]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Endovascular Thrombectomy Plus Medical Management | Medical Management
All-Cause Mortality (participants affected / at risk) | 68/178 | 71/174
Serious Adverse Events (participants affected / at risk) | 129/178 | 123/174
Other Adverse Events (participants affected / at risk) | 77/178 | 59/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Thrombectomy Plus Medical Management (N=178) | Medical Management (N=174)
Access Site Complication - Arterial Occlusion (Vascular disorders) | 3 | 0
Access Site Complication - Hematoma (Vascular disorders) | 1 | 0
Access Site Complication - Infection (Vascular disorders) | 1 | 0
Acute Arterial Occlusion (Acute Limb Ischemia) (Vascular disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 9 | 9
Cerebral Edema with Midline Shift (Nervous system disorders) | 64 | 57
Cerebritis (Nervous system disorders) | 1 | 0
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Deep Vein Thrombosis (Vascular disorders) | 2 | 2
Delirium, Cognitive Dysfunction (Nervous system disorders) | 9 | 5
Endocarditis (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 7 | 8
Hyperglycemic Hyperosmolar State (Endocrine disorders) | 0 | 1
Lower respiratory infection (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 18 | 21
Myocardial infarction (Cardiac disorders) | 2 | 3
Neurological Deterioration (Nervous system disorders) | 44 | 27
New Stroke (Nervous system disorders) | 6 | 5
Pericardial effusion (Cardiac disorders) | 1 | 0
Progression of Disease, Palliative Care Decision (Nervous system disorders) | 25 | 31
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory failure (Reproductive system and breast disorders) | 30 | 19
Sepsis, Systemic inflammatory response syndrome (Infections and infestations) | 11 | 9
Symptomatic Intracranial Hemorrhage (Nervous system disorders) | 1 | 2
Urinary Tract Infection (Renal and urinary disorders) | 12 | 13
Wound Infection (Skin and subcutaneous tissue disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Thrombectomy Plus Medical Management (N=178) | Medical Management (N=174)
Alcohol Withdrawal (General disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 4
Anxiety (Psychiatric disorders) | 0 | 1
Asymptomatic Intracranial Hemorrhage (Nervous system disorders) | 0 | 1
Cardiac Arrythmia (Cardiac disorders) | 21 | 20
Carotid Cavernous Fistula (Nervous system disorders) | 1 | 0
Cerebral Vasospasm (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 0
Diaphoresis (General disorders) | 1 | 1
Dizziness (General disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Epidural Hemorrhage (Nervous system disorders) | 0 | 1
Epistaxis (Vascular disorders) | 2 | 0
Evolution of infarction on the brain imaging (Nervous system disorders) | 8 | 8
Eye Complications (Eye disorders) | 2 | 0
Fall (General disorders) | 2 | 4
Fever (General disorders) | 7 | 9
Gastrointestinal Complications (Gastrointestinal disorders) | 19 | 8
Hallucination (Cardiac disorders) | 1 | 0
Headache (General disorders) | 9 | 2
Hematoma (Vascular disorders) | 2 | 1
Hypertension (Cardiac disorders) | 1 | 3
Hypotension (Cardiac disorders) | 4 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Insomnia (General disorders) | 3 | 0
Lactose intolerance reaction (Gastrointestinal disorders) | 1 | 0
Laryngeal Edema (Immune system disorders) | 1 | 0
Lethargy (General disorders) | 4 | 4
Liver Injury (Hepatobiliary disorders) | 5 | 1
Musculoskeletal Complications (Musculoskeletal and connective tissue disorders) | 9 | 6
Nausea (General disorders) | 4 | 2
near syncopal episode (Cardiac disorders) | 1 | 0
Non-Cerebral Thrombotic Events (Vascular disorders) | 5 | 1
ocular nerve damage (Eye disorders) | 1 | 0
Other Renal Complications (Renal and urinary disorders) | 14 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Progression of Disease (Nervous system disorders) | 16 | 11
SDH (Nervous system disorders) | 1 | 0
Seizures (Nervous system disorders) | 2 | 2
Skin Complications (Skin and subcutaneous tissue disorders) | 10 | 1
Splenic infarct (Blood and lymphatic system disorders) | 1 | 0
Stent Thrombosis (Vascular disorders) | 1 | 0
Symptomatic Carotid Artery Stenosis (Vascular disorders) | 0 | 1
Syndrome of inappropriate ADH production (Endocrine disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tremors (Nervous system disorders) | 0 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vessel dissection (Nervous system disorders) | 4 | 0
Vessel perforation (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT03876457/Prot_SAP_000.pdf